CLINICAL TRIAL: NCT00347360
Title: A Randomized, Double-Blind, Double-Dummy, Parallel Group, Factorial Design Trial to Assess the Efficacy and Safety of up to Six Weeks Treatment With 20mg, 40mg, or 80mg QD Doses of Carvedilol Controlled Release Formulation (COREG CR) or 10mg, 20mg, or 40mg QD Doses of Lisinopril (Zestril) or a Combination of One of the Doses of Each Medication
Brief Title: The COREG And Lisinopril Combination Therapy In Hypertensive Subjects (COSMOS) Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFD105453
Record Dates: First submitted 2006-06-29; First posted 2006-07-04 (Estimated); Results first posted 2009-11-09 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: carvedilol; hypertension; lisinopril; factorial
MeSH Terms: conditions — Hypertension | interventions — Lisinopril

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- lisinopril (Experimental): lisinopril
  Interventions: Drug: lisinopril
- carvedilol (Experimental): carvedilol controlled release formulation
  Interventions: Drug: carvedilol controlled release formulation

INTERVENTIONS:
Drug: lisinopril
  Arms: lisinopril
Drug: carvedilol controlled release formulation
  Other Names: lisinopril
  Arms: carvedilol

SUMMARY:
This is a randomized, double-blind, double-dummy, parallel group trial employing 15 cells of a 4x4 factorial design (no placebo)to compare the hypertensive effects in patients with Stage 1 and Stage 2 hypertension of carvedilol (20, 40 or 80 mg daily) alone, lisinopril (10, 20 or 40 mg daily) alone, and all combinations of the doses.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Double-Dummy, Parallel Group, Factorial Design Trial to Assess the Efficacy and Safety of up to Six Weeks Treatment with 20mg, 40mg, or 80mg QD Doses of Carvedilol Controlled Release Formulation (COREG CR) or 10mg, 20mg, or 40mg QD Doses of Lisinopril (ZESTRIL) or a Combination of One of the Doses of Each Medication

ELIGIBILITY:
Inclusion Criteria:

* Subject has given signed informed consent.
* Subject is male or female 18 years of age at the time informed consent is signed.
* At the Screening visit, subject has a documented history or current presentation with stage 1 or stage 2 hypertension (see Section 15.1, Appendix 1 and Section 15.4, Appendix 4) which meets one of the following criteria. Note: All blood pressures are mean sitting cuff pressures:

Documented history of hypertension and receiving two antihypertensive medications with mean sDBP <90 mmHg or for diabetic subjects (defined as having an established diagnosis of diabetes or receiving treatment for diabetes), mean sDBP <80 mmHg. Subjects taking beta blockers, clonidine, or other antihypertensive medications where abrupt discontinuation would be of clinical concern must be tapered off the medication during the Washout/Placebo Run-in phase to avoid rebound hypertension. All subjects must be able to be safely withdrawn from all antihypertensive treatment during the Washout/Placebo Run-in phase. Subjects should not be enrolled if the investigator thinks it is likely the subject's mean sDBP will exceed 109 mmHg or their mean sSBP will exceed 180 mmHg during the Washout/Placebo Run-in phase (NOTE: A combination drug containing two antihypertensive agents represents two antihypertensive medications [e.g., Hyzaar is losartan potassium AND hydrochlorothiazide, therefore, counts as two antihypertensive medications].) OR Receiving one antihypertensive medication with mean sDBP =109 mmHg and can be safely withdrawn from all antihypertensive medication during the Washout/Placebo Run-in phase. Any subject who is receiving beta-blockers, clonidine, or other antihypertensive medications where abrupt discontinuation would be of clinical concern must have the dose tapered down during the Washout/Placebo Run-in phase to avoid rebound hypertension. All subjects must be able to be safely withdrawn from all antihypertensive treatment during the Washout/Placebo Run-in phase. Subjects should not be enrolled if the investigator thinks it is likely the subject's mean sDBP will exceed 109 mmHg or their mean sSBP will exceed 180 mmHg during the Washout/Placebo Run-in phase.

(NOTE: A combination drug containing two antihypertensive agents represents two antihypertensive medications [e.g., Hyzaar is losartan potassium AND hydrochlorothiazide, therefore, counts as two antihypertensive medications].

OR Untreated/newly diagnosed subjects: mean sDBP =95 and =109, or for diabetic subjects, mean sDBP =85 and =109 (see Section 15.1, Appendix 1). If newly diagnosed, must have qualifying blood pressure confirmed on two consecutive visits with the mean sDBP value not differing more than 8 mmHg. (Previously untreated subjects include subjects who have not been treated for hypertension in the last two months.).

* At Baseline:

DAY BEFORE RANDOMIZATION: Prior to having the baseline ABPM equipment placed, subject has mean sitting cuff DBP that is ≥93 and ≤111 mmHg (or for diabetic subjects, ≥83 and ≤111 mmHg). Subjects who were taking antihypertensive medication at Screening and do not meet this criterion after one week (or 5 half-lives, whichever is longer), can return in one week ±1day and have his/her blood pressure evaluated again for this inclusion criterion.

AND

RANDOMIZATON DAY: After completion of the ABPM assessment, subject meets the following ABPM (both 12 hr and 24 hr) criteria (see Section 15.1, Appendix 1):

* Mean 12-hour daytime (9 AM to 9 PM) DBP ≥90 and ≤109mmHg (or for diabetic subjects, ≥80 and ≤109mmHg)
* At least 75% of the programmed readings properly recorded over 24-hour monitoring period
* No more than two non-consecutive hours with less than two successful readings per hour while awake, and no more than two consecutive hours with less than one successful reading per hour during the sleep period over the 24-hour monitoring period
* At least two successful readings per hour for three of the last four hours of recording (trough period i.e., 20-24 hour during which subjects must be awake) with a total of at least 7 successful readings over this period.

Exclusion Criteria:

* Subject is taking ≥3 antihypertensive medications. (NOTE: A combination drug containing two antihypertensive agents represents two antihypertensive medications [e.g., Hyzaar is losartan potassium AND hydrochlorothiazide, therefore, counts as two antihypertensive medications].)
* Subject has DBP =90 mmHg (or for diabetic subjects, DBP =80 mmHg) on two antihypertensive medications.
* Subject has any known contraindication to ACE inhibitors (e.g., ACE-induced cough, angioedema or negative renal effects), or blocker treatment.
* Hyperkalemia or history of hyperkalemia resulting from either Type IV RTA (renal tubular acidosis) or previous ACEi therapy.
* Is female of childbearing potential. NOTE: Female subjects who are postmenopausal (i.e., no menstrual period for a minimum of 12 months prior to Screening) or surgically sterilized are eligible for the study. If judged appropriate, a postmenopausal woman may be required to have a documented negative urine pregnancy test.
* Subject has malignant (accelerated) hypertension, history of malignant hypertension, or secondary forms of hypertension.
* Subject has mean sitting SBP =180 mmHg.
* Subject has advanced hypertensive retinopathy (Keith Wagner Grade IV).
* Subject has Type 1 diabetes mellitus, or those with Type 2 having HbA1c ≥9% at Screening.
* Subject has uncorrected primary obstructive or severe regurgitative valvular disease, nondilated (restrictive) or hypertrophic cardiomyopathies.
* Subject has any of the following conditions:

uncontrollable or symptomatic arrhythmias unstable angina or angina treated with a beta-blocker sick sinus syndrome or second or third degree heart block (unless treated with a permanent, functioning pacemaker) bradycardia (sitting heart rate <55 bpm) history of myocardial infarction stroke within 3 months of Screening

* Subject is in atrial fibrillation.
* Subject has Congestive Heart Failure NYHA (New York Heart Association) class II-IV [The Criteria Committee of the New York Heart Association, 1994].
* Current clinical evidence of asthma or chronic obstructive pulmonary disease (e.g., severe emphysema or chronic bronchitis) requiring long term use of inhaled oral bronchodilator or steroid drug therapy; also subjects with a history of bronchospastic disease not undergoing active therapy in whom, in the investigator's opinion, treatment with the study medication could provoke bronchospasm; or requirement for or anticipated treatment with beta-2 agonist therapy (e.g., albuterol [Ventolin, Proventil], metaproterenol [Alupent], pirbuterol [Maxair], terbutaline [Brethaire], isoetharine [Bronkosol], and Levalbuterol [Xopenex]).
* Subject has evidence of any of the following clinically significant diseases that could impair the absorption, metabolism, or excretion of orally-administered medication:

renal disease defined as estimated Glomerular Filtration Rate (eGFR) <30mL/min per 1.73 m2 hepatic disease (i.e., ALT or AST levels greater than three times the upper limit of normal range, history of hepatic impairment, or by clinical assessment) chronic biliary disorders gastric bypass surgery

* Subject has endocrine disorders that affect blood pressure (e.g., pheochromocytoma, active and untreated hypo- or hyperthyroidism).
* Subject has systemic disease, including cancer, with reduced (<12 months) life expectancy.
* Subject has used an investigational drug within 30 days or 5 half-lives (whichever is longer) preceding Screening.
* Subject has a history of a psychological illness/condition that would interfere with their ability to understand or complete the requirements of the study.
* Subject has any condition that, in the opinion of the Investigator and/or the GSK Medical Monitor, places the subject at an unacceptable risk as a participant in this trial.
* Subject is receiving ongoing treatment or is anticipated to receive treatment with any of the following medications during treatment with double blind study medication:

any antihypertensive medication except for assigned study medication. This would include alpha blockers or other medications that may be used to treat hypertension and other conditions unrelated to hypertension; monoamine oxidase (MAO) inhibitors; any Class I or III antiarrhythmic; beta-2-agonists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 654 (Actual)
Dates: Start 2006-07; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (134):
- United States (134):
  - GSK Investigational Site, Anniston, Alabama
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Haleyville, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Muscle Shoals, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Phoenix, Arizona, Arizona
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Sun City, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Searcy, Arkansas
  - GSK Investigational Site, Beuna Park, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Carlsbad, California
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Loma Linda, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Pico Rivera, California
  - GSK Investigational Site, Rancho Cordova, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Walnut Creek, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Wilmington, Delaware
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Jacksonville Beach, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Palm Harbor, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Gainesville, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Sandersville, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Aurora, Illinois
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Melrose Park, Illinois
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Bloomington, Indiana
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Ames, Iowa
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Slidell, Louisiana
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Taunton, Massachusetts
  - GSK Investigational Site, Bingham Farms, Michigan
  - GSK Investigational Site, Brooklyn Center, Minnesota
  - GSK Investigational Site, Missoula, Montana
  - GSK Investigational Site, O Fallon, Montana
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Cherry Hill, New Jersey
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Ridgewood, New Jersey
  - GSK Investigational Site, Voorhees Township, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Kingston, New York
  - GSK Investigational Site, Lewinston, New York
  - GSK Investigational Site, Tonawanda, New York
  - GSK Investigational Site, Asheville, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, High Point, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Fargo, North Dakota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Beaver, Pennsylvania
  - GSK Investigational Site, Doylestown, Pennsylvania
  - GSK Investigational Site, Erie, Pennsylvania
  - GSK Investigational Site, Havertown, Pennsylvania
  - GSK Investigational Site, Landsdale, Pennsylvania
  - GSK Investigational Site, Leetsdale, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Warminster, Pennsylvania
  - GSK Investigational Site, West Chester, Pennsylvania
  - GSK Investigational Site, Beaufort, South Carolina
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Hilton Head Island, South Carolina
  - GSK Investigational Site, Manning, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Sumter, South Carolina
  - GSK Investigational Site, Taylors, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Jackson, Tennessee
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Selmer, Tennessee
  - GSK Investigational Site, Arlington, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Georgetown, Texas
  - GSK Investigational Site, Grand Prairie/Texas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Longview, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Sugar Land, Texas
  - GSK Investigational Site, Temple, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Murray, Utah
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Sandy City, Utah
  - GSK Investigational Site, Arlington, Virginia
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Chester, Virginia
  - GSK Investigational Site, Fairfax, Virginia
  - GSK Investigational Site, Manassas, Virginia
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Tacoma, Washington
  - GSK Investigational Site, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Bakris GL, Iyengar M, Lukas MA, Ordronneau P, Weber MA. Effect of combining extended-release carvedilol and lisinopril in hypertension: results of the COSMOS study. J Clin Hypertens (Greenwich). 2010 Sep;12(9):678-86. doi: 10.1111/j.1751-7176.2010.00341.x. Epub 2010 Jul 8. PMID 20883227
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: CFD105453 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: CFD105453 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: CFD105453 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: CFD105453 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: CFD105453 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: CFD105453 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: CFD105453 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Lisinopril 10: lisinopril 10 milligrams (mg) once daily
- Lisinopril 20: lisinopril 20 mg once daily
- Lisinopril 40: lisinopril 40 mg once daily
- Carvedilol Controlled Release 20: carvedilol controlled release (CR) 20 mg once daily
- Carvedilol Controlled Release 40: carvedilol CR 40 mg once daily
- Carvedilol Controlled Release 80: carvedilol CR 80 mg once daily
- Carvedilol Controlled Release 20 Lisinopril 10: carvedilol CR 20 mg plus lisinopril 10 mg once daily
- Carvedilol Controlled Release 20 Lisinopril 20: carvedilol CR 20 mg plus lisinopril 20 mg once daily
- Carvedilol Controlled Release 20 Lisinopril 40: carvedilol CR 20 mg plus lisinopril 40 mg once daily
- Carvedilol Controlled Release 40 Lisinopril 10: carvedilol CR 40 mg plus lisinopril 10 mg once daily
- Carvedilol Controlled Release 40 Lisinopril 20: carvedilol CR 40 mg plus lisinopril 20 mg once daily
- Carvedilol Controlled Release 40 Lisinopril 40: carvedilol CR 40 mg plus lisinopril 40 mg once daily
- Carvedilol Controlled Release 80 Lisinopril 10: carvedilol CR 80 mg plus lisinopril 10 mg once daily
- Carvedilol Controlled Release 80 Lisinopril 20: carvedilol CR 80 mg plus lisinopril 20 mg once daily
- Carvedilol Controlled Release 80 Lisinopril 40: carvedilol CR 80 mg plus lisinopril 40 mg once daily
Period: Overall Study
Arm/Group | Lisinopril 10 | Lisinopril 20 | Lisinopril 40 | Carvedilol Controlled Release 20 | Carvedilol Controlled Release 40 | Carvedilol Controlled Release 80 | Carvedilol Controlled Release 20 Lisinopril 10 | Carvedilol Controlled Release 20 Lisinopril 20 | Carvedilol Controlled Release 20 Lisinopril 40 | Carvedilol Controlled Release 40 Lisinopril 10 | Carvedilol Controlled Release 40 Lisinopril 20 | Carvedilol Controlled Release 40 Lisinopril 40 | Carvedilol Controlled Release 80 Lisinopril 10 | Carvedilol Controlled Release 80 Lisinopril 20 | Carvedilol Controlled Release 80 Lisinopril 40
Started | 44 | 43 | 43 | 43 | 44 | 44 | 44 | 43 | 44 | 44 | 44 | 43 | 44 | 44 | 43
Completed | 39 | 35 | 37 | 30 | 39 | 36 | 37 | 40 | 38 | 35 | 39 | 37 | 34 | 36 | 39
Not Completed | 5 | 8 | 6 | 13 | 5 | 8 | 7 | 3 | 6 | 9 | 5 | 6 | 10 | 8 | 4
Not completed — Adverse Event | 1 | 2 | 0 | 4 | 1 | 2 | 2 | 0 | 2 | 3 | 3 | 1 | 3 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 3 | 1 | 2 | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 4 | 1 | 2 | 1 | 1 | 1 | 1 | 0 | 3 | 4 | 2 | 1
Not completed — Lack of Efficacy | 1 | 1 | 3 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Reason not listed/blank | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Per sponsors instruction | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — P.I. recommended due to blood pressure | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Subject did not meet end of study ABPM | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Abnormal lab values | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — PI recommended early withdrawal | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Did not meet criteria before ABPM | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Randomized in error | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Failed inclusion criteria #4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Prolonged duration between visits | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Subject left town, ran out of study drug | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Subject refuse to sign updated consent | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Visits conflicted with new job | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lisinopril 10 | Lisinopril 20 | Lisinopril 40 | Carvedilol Controlled Release 20 | Carvedilol Controlled Release 40 | Carvedilol Controlled Release 80 | Carvedilol Controlled Release 20 Lisinopril 10 | Carvedilol Controlled Release 20 Lisinopril 20 | Carvedilol Controlled Release 20 Lisinopril 40 | Carvedilol Controlled Release 40 Lisinopril 10 | Carvedilol Controlled Release 40 Lisinopril 20 | Carvedilol Controlled Release 40 Lisinopril 40 | Carvedilol Controlled Release 80 Lisinopril 10 | Carvedilol Controlled Release 80 Lisinopril 20 | Carvedilol Controlled Release 80 Lisinopril 40 | Total
Number analyzed (Participants) | 44 | 43 | 43 | 43 | 44 | 44 | 44 | 43 | 44 | 44 | 44 | 43 | 44 | 44 | 43 | 654
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.3 (10.53) | 53.3 (10.69) | 51.1 (10.70) | 53.2 (9.41) | 54.1 (10.94) | 54.3 (8.64) | 53.3 (9.60) | 55.5 (8.39) | 53.5 (10.51) | 51.9 (9.08) | 51.5 (9.32) | 57.9 (9.27) | 52.5 (11.11) | 50.9 (9.51) | 51.5 (8.69) | 53.1 (9.86)
Gender [Count of Participants; unit: Participants]
  Female | 17 | 17 | 15 | 20 | 12 | 19 | 13 | 18 | 14 | 13 | 13 | 18 | 15 | 14 | 14 | 232
  Male | 27 | 26 | 28 | 23 | 32 | 25 | 31 | 25 | 30 | 31 | 31 | 25 | 29 | 30 | 29 | 422
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 10 | 14 | 9 | 16 | 11 | 13 | 12 | 11 | 12 | 18 | 14 | 13 | 16 | 14 | 11 | 194
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
  Asian | 3 | 1 | 3 | 1 | 2 | 2 | 2 | 1 | 2 | 2 | 3 | 1 | 3 | 3 | 4 | 33
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 29 | 28 | 31 | 26 | 30 | 29 | 30 | 30 | 29 | 23 | 27 | 27 | 25 | 26 | 27 | 417
  Race not provided by patient | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 6 in 24 Hour (hr) Mean Diastolic Blood Pressure
Description: Ambulatory blood pressure monitoring (ABPM) was completed at Baseline and at the end of treatment/Week 6 or early withdrawal by standard electronic ABPM equipment worn by the subject for 24-hr of ambulatory activity. The 24 hr assessment period started at the time of the first reading and ended exactly 24 hr later on the following day. Data collected included mean diastolic blood pressure (DBP).
Time Frame: Baseline, Week 6.
Population: ABPM Population with Last Observation Carried Forward (LOCF): This comprised all randomized subjects with efficacy (vital signs) data after a minimum of 2 weeks on treatment with valid Baseline and on-therapy ABPM measures. All efficacy data derived from ABPM assessments were summarized by this population.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lisinopril 10 | Lisinopril 20 | Lisinopril 40 | Carvedilol Controlled Release 20 | Carvedilol Controlled Release 40 | Carvedilol Controlled Release 80 | Carvedilol Controlled Release 20 Lisinopril 10 | Carvedilol Controlled Release 20 Lisinopril 20 | Carvedilol Controlled Release 20 Lisinopril 40 | Carvedilol Controlled Release 40 Lisinopril 10 | Carvedilol Controlled Release 40 Lisinopril 20 | Carvedilol Controlled Release 40 Lisinopril 40 | Carvedilol Controlled Release 80 Lisinopril 10 | Carvedilol Controlled Release 80 Lisinopril 20 | Carvedilol Controlled Release 80 Lisinopril 40
Number analyzed (Participants) | 29 | 30 | 38 | 27 | 34 | 33 | 35 | 37 | 34 | 32 | 35 | 34 | 28 | 33 | 34
mmHg | -5.79 (5.922) | -8.11 (8.811) | -7.37 (5.914) | -4.40 (5.182) | -7.61 (4.880) | -6.52 (6.408) | -9.29 (7.226) | -8.57 (6.585) | -10.19 (6.899) | -9.36 (7.426) | -10.96 (8.388) | -10.37 (7.234) | -10.93 (5.517) | -11.09 (8.719) | -11.92 (6.887)
Statistical Analysis 1: Comparison: Lisinopril 10 vs Lisinopril 20 vs Lisinopril 40 vs Carvedilol Controlled Release 20 vs Carvedilol Controlled Release 40 vs Carvedilol Controlled Release 80 vs Carvedilol Controlled Release 20 Lisinopril 10 vs Carvedilol Controlled Release 20 Lisinopril 20 vs Carvedilol Controlled Release 20 Lisinopril 40 vs Carvedilol Controlled Release 40 Lisinopril 10 vs Carvedilol Controlled Release 40 Lisinopril 20 vs Carvedilol Controlled Release 40 Lisinopril 40 vs Carvedilol Controlled Release 80 Lisinopril 10 vs Carvedilol Controlled Release 80 Lisinopril 20 vs Carvedilol Controlled Release 80 Lisinopril 40; This is an omnibus test to investigate the existence of at least one combination dose that outperforms its components; Test type: Superiority or Other; p > 0.1, Hung AVE test, see comments; Hung AVE Test Statistic: -0.41499. Tests an average of the minimum gains (in response) for the 9 combination cells over corresponding monotherapies

2. Primary Outcome: Change From Baseline to Week 6 in Trough Diastolic Blood Pressure
Description: Trough ABPM was the average across 20-24 hr after dosing for each subject.
Time Frame: Baseline, Week 6
Population: ABPM Population with LOCF: This comprised all randomized subjects with efficacy (vital signs) data after a minimum of 2 weeks on treatment with valid Baseline and on-therapy ABPM measures. All efficacy data derived from ABPM assessments were summarized by this population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lisinopril 10 | Lisinopril 20 | Lisinopril 40 | Carvedilol Controlled Release 20 | Carvedilol Controlled Release 40 | Carvedilol Controlled Release 80 | Carvedilol Controlled Release 20 Lisinopril 10 | Carvedilol Controlled Release 20 Lisinopril 20 | Carvedilol Controlled Release 20 Lisinopril 40 | Carvedilol Controlled Release 40 Lisinopril 10 | Carvedilol Controlled Release 40 Lisinopril 20 | Carvedilol Controlled Release 40 Lisinopril 40 | Carvedilol Controlled Release 80 Lisinopril 10 | Carvedilol Controlled Release 80 Lisinopril 20 | Carvedilol Controlled Release 80 Lisinopril 40
Number analyzed (Participants) | 29 | 29 | 38 | 27 | 34 | 33 | 33 | 35 | 34 | 29 | 33 | 33 | 28 | 33 | 34
mmHg | -6.40 (7.982) | -6.08 (8.735) | -8.16 (7.299) | -2.34 (7.060) | -7.76 (8.285) | -5.26 (9.530) | -5.14 (7.002) | -6.36 (9.080) | -7.22 (11.284) | -6.79 (9.210) | -7.76 (11.202) | -4.90 (8.508) | -6.54 (8.305) | -7.26 (9.345) | -8.42 (7.903)
Statistical Analysis 1: Comparison: Lisinopril 10 vs Lisinopril 20 vs Lisinopril 40 vs Carvedilol Controlled Release 20 vs Carvedilol Controlled Release 40 vs Carvedilol Controlled Release 80 vs Carvedilol Controlled Release 20 Lisinopril 10 vs Carvedilol Controlled Release 20 Lisinopril 20 vs Carvedilol Controlled Release 20 Lisinopril 40 vs Carvedilol Controlled Release 40 Lisinopril 10 vs Carvedilol Controlled Release 40 Lisinopril 20 vs Carvedilol Controlled Release 40 Lisinopril 40 vs Carvedilol Controlled Release 80 Lisinopril 10 vs Carvedilol Controlled Release 80 Lisinopril 20 vs Carvedilol Controlled Release 80 Lisinopril 40; This is an omnibus test to investigate the existence of at least one combination dose that outperforms its components; Test type: Superiority or Other; p > 0.1, Hung AVE test, see comments; Hung AVE Test Statistic: -0.00485. Tests an average of the minimum gains (in response) for the 9 combination cells over corresponding monotherapies

3. Secondary Outcome: Change From Baseline to Week 6 in 24 Hour Mean Systolic Blood Pressure
Description: Ambulatory blood pressure monitoring (ABPM) was completed at Baseline and at the end of treatment/Week 6 or early withdrawal by standard electronic ABPM equipment worn by the subject for 24-hr of ambulatory activity. The 24 hr assessment period started at the time of the first reading and ended exactly 24 hr later on the following day. Data collected included mean systolic blood pressure (SBP).
Time Frame: Baseline, Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lisinopril 10 | Lisinopril 20 | Lisinopril 40 | Carvedilol Controlled Release 20 | Carvedilol Controlled Release 40 | Carvedilol Controlled Release 80 | Carvedilol Controlled Release 20 Lisinopril 10 | Carvedilol Controlled Release 20 Lisinopril 20 | Carvedilol Controlled Release 20 Lisinopril 40 | Carvedilol Controlled Release 40 Lisinopril 10 | Carvedilol Controlled Release 40 Lisinopril 20 | Carvedilol Controlled Release 40 Lisinopril 40 | Carvedilol Controlled Release 80 Lisinopril 10 | Carvedilol Controlled Release 80 Lisinopril 20 | Carvedilol Controlled Release 80 Lisinopril 40
Number analyzed (Participants) | 29 | 30 | 38 | 27 | 34 | 33 | 35 | 37 | 34 | 32 | 35 | 34 | 28 | 33 | 34
mmHg | -9.19 (9.415) | -13.58 (16.429) | -10.60 (8.842) | -6.15 (6.887) | -9.84 (8.471) | -10.38 (8.204) | -12.06 (11.058) | -11.58 (11.112) | -14.16 (10.783) | -11.68 (10.218) | -14.03 (11.954) | -13.90 (10.237) | -15.60 (9.777) | -15.93 (12.501) | -15.59 (11.055)

4. Secondary Outcome: Change From Baseline to Week 6 in Trough Systolic Blood Pressure
Description: Trough ABPM was the average across 20-24 hr after dosing for each subject.
Time Frame: Baseline, Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lisinopril 10 | Lisinopril 20 | Lisinopril 40 | Carvedilol Controlled Release 20 | Carvedilol Controlled Release 40 | Carvedilol Controlled Release 80 | Carvedilol Controlled Release 20 Lisinopril 10 | Carvedilol Controlled Release 20 Lisinopril 20 | Carvedilol Controlled Release 20 Lisinopril 40 | Carvedilol Controlled Release 40 Lisinopril 10 | Carvedilol Controlled Release 40 Lisinopril 20 | Carvedilol Controlled Release 40 Lisinopril 40 | Carvedilol Controlled Release 80 Lisinopril 10 | Carvedilol Controlled Release 80 Lisinopril 20 | Carvedilol Controlled Release 80 Lisinopril 40
Number analyzed (Participants) | 29 | 29 | 38 | 27 | 34 | 33 | 33 | 35 | 34 | 29 | 33 | 33 | 28 | 33 | 34
mmHg | -9.47 (13.301) | -7.52 (12.221) | -9.54 (9.968) | -0.96 (11.447) | -9.27 (12.362) | -5.68 (14.539) | -6.44 (9.739) | -9.27 (13.582) | -9.88 (14.356) | -8.87 (11.954) | -8.11 (13.732) | -5.82 (13.878) | -9.80 (11.196) | -10.74 (12.813) | -10.00 (12.091)

5. Secondary Outcome: Dose-response Treatment Estimates: Change From Baseline to Week 6 in 24 Hour Mean DBP by ABPM (Ambulatory Blood Pressure Monitoring)
Description: Evaluation of the dose-response relationship between incremental doses of carvedilol CR and lisinopril and mean 24-hr ABPM DBP.
Time Frame: Baseline, Week 6
Population: as for outcome 2
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Lisinopril 10 | Lisinopril 20 | Lisinopril 40 | Carvedilol Controlled Release 20 | Carvedilol Controlled Release 40 | Carvedilol Controlled Release 80 | Carvedilol Controlled Release 20 Lisinopril 10 | Carvedilol Controlled Release 20 Lisinopril 20 | Carvedilol Controlled Release 20 Lisinopril 40 | Carvedilol Controlled Release 40 Lisinopril 10 | Carvedilol Controlled Release 40 Lisinopril 20 | Carvedilol Controlled Release 40 Lisinopril 40 | Carvedilol Controlled Release 80 Lisinopril 10 | Carvedilol Controlled Release 80 Lisinopril 20 | Carvedilol Controlled Release 80 Lisinopril 40
Number analyzed (Participants) | 29 | 30 | 38 | 27 | 34 | 33 | 35 | 37 | 34 | 32 | 35 | 34 | 28 | 33 | 34
mmHg | -5.77 (0.821) | -7.55 (0.717) | -7.49 (0.877) | -5.11 (0.821) | -6.61 (0.718) | -7.13 (0.925) | -8.08 (0.472) | -9.83 (0.536) | -9.71 (0.657) | -9.55 (0.534) | -11.3 (0.645) | -11.1 (0.702) | -10.0 (0.696) | -11.7 (0.722) | -11.4 (1.042)

6. Secondary Outcome: Change From Baseline to Week 6 in Trough to Peak Ratios of DBP by 24 Hour ABPM (Ambulatory Blood Pressure Monitoring)
Description: Trough (20-24 hr) to peak (3-7 hr) ratios of DBP were examined in order to evaluate the extent to which once-daily criteria were met (ie trough:peak > 50%). Trough to peak ratios were calculated from change trough mean/change peak mean x 100.
Time Frame: Baseline, Week 6
Population: as for outcome 2
Measure: Number; unit: trough:peak ratio x 100%
Arm/Group | Lisinopril 10 | Lisinopril 20 | Lisinopril 40 | Carvedilol Controlled Release 20 | Carvedilol Controlled Release 40 | Carvedilol Controlled Release 80 | Carvedilol Controlled Release 20 Lisinopril 10 | Carvedilol Controlled Release 20 Lisinopril 20 | Carvedilol Controlled Release 20 Lisinopril 40 | Carvedilol Controlled Release 40 Lisinopril 10 | Carvedilol Controlled Release 40 Lisinopril 20 | Carvedilol Controlled Release 40 Lisinopril 40 | Carvedilol Controlled Release 80 Lisinopril 10 | Carvedilol Controlled Release 80 Lisinopril 20 | Carvedilol Controlled Release 80 Lisinopril 40
Number analyzed (Participants) | 29 | 29 | 38 | 27 | 34 | 33 | 33 | 35 | 34 | 29 | 33 | 34 | 28 | 33 | 34
trough:peak ratio x 100% | 133.33 | 61.04 | 114.45 | 34.11 | 71.00 | 49.67 | 44.50 | 49.46 | 59.47 | 54.71 | 52.86 | 37.93 | 41.95 | 53.54 | 52.07

7. Secondary Outcome: Overall Description of Safety in Each Treatment Group Using Adverse Events, Laboratory Evaluations, ECG Changes, Vital Sign Changes, and Withdrawal Rates.
Description: Refer to Adverse Event section for safety information.
Time Frame: Weeks 1 through 48
Reporting Status: Not Posted

8. Secondary Outcome: Change From Baseline to Week 6 in Mean SBP and DBP Measured in Morning by 24 Hour ABPM
Description: Mean changes from Baseline to Week 6 in DBP and SBP measured by 24hr ABPM at the end of up-titration recorded in the morning. The morning assessment period started at or after 6 am and ended immediately before 12 noon.
Time Frame: Morning BP, Baseline, Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lisinopril 10 | Lisinopril 20 | Lisinopril 40 | Carvedilol Controlled Release 20 | Carvedilol Controlled Release 40 | Carvedilol Controlled Release 80 | Carvedilol Controlled Release 20 Lisinopril 10 | Carvedilol Controlled Release 20 Lisinopril 20 | Carvedilol Controlled Release 20 Lisinopril 40 | Carvedilol Controlled Release 40 Lisinopril 10 | Carvedilol Controlled Release 40 Lisinopril 20 | Carvedilol Controlled Release 40 Lisinopril 40 | Carvedilol Controlled Release 80 Lisinopril 10 | Carvedilol Controlled Release 80 Lisinopril 20 | Carvedilol Controlled Release 80 Lisinopril 40
Number analyzed (Participants) | 29 | 30 | 38 | 27 | 34 | 32 | 35 | 37 | 34 | 32 | 35 | 34 | 28 | 33 | 34
mmHg
  Change in Morning SBP from Baseline to Week 6 | -9.37 (9.564) | -14.53 (17.166) | -10.76 (9.112) | -6.23 (9.159) | -10.42 (8.815) | -13.70 (10.056) | -13.89 (12.288) | -10.22 (12.734) | -14.50 (12.031) | -12.78 (14.700) | -14.29 (14.136) | -14.84 (13.383) | -17.09 (13.194) | -14.52 (15.111) | -17.12 (14.016)
  Change in Morning DBP from Baseline to Week 6 | -6.12 (8.457) | -9.20 (10.516) | -7.62 (8.033) | -5.01 (7.141) | -6.82 (6.279) | -7.53 (8.206) | -9.21 (9.474) | -7.86 (8.416) | -10.04 (8.489) | -8.79 (10.902) | -11.15 (10.411) | -9.96 (10.730) | -11.95 (8.060) | -10.71 (11.012) | -12.46 (8.763)

9. Secondary Outcome: Change From Baseline to Week 6 in Mean SBP and DBP Measured in Afternoon by 24hr ABPM
Description: Mean changes from Baseline to Week 6 in SBP and DBP measured by 24hr ABPM at the end of up-titration recorded in the afternoon. The afternoon assessment period started at or after 12 noon and ended immediately before 6 pm.
Time Frame: Afternoon BP, Baseline, Week 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lisinopril 10 | Lisinopril 20 | Lisinopril 40 | Carvedilol Controlled Release 20 | Carvedilol Controlled Release 40 | Carvedilol Controlled Release 80 | Carvedilol Controlled Release 20 Lisinopril 10 | Carvedilol Controlled Release 20 Lisinopril 20 | Carvedilol Controlled Release 20 Lisinopril 40 | Carvedilol Controlled Release 40 Lisinopril 10 | Carvedilol Controlled Release 40 Lisinopril 20 | Carvedilol Controlled Release 40 Lisinopril 40 | Carvedilol Controlled Release 80 Lisinopril 10 | Carvedilol Controlled Release 80 Lisinopril 20 | Carvedilol Controlled Release 80 Lisinopril 40
Number analyzed (Participants) | 29 | 30 | 38 | 27 | 34 | 33 | 35 | 37 | 34 | 32 | 35 | 34 | 28 | 33 | 34
mmHg
  Change in Afternoon SBP from Baseline to Week 6 | -9.68 (11.399) | -17.21 (19.772) | -10.53 (13.359) | -9.69 (10.094) | -13.34 (9.669) | -13.76 (11.796) | -13.96 (13.128) | -15.54 (13.503) | -16.38 (13.285) | -14.51 (13.433) | -17.97 (14.622) | -17.82 (13.042) | -20.91 (13.704) | -20.46 (17.611) | -19.36 (14.893)
  Change in Afternoon DBP from Baseline to Week 6 | -5.62 (7.969) | -10.25 (12.250) | -6.67 (7.800) | -6.27 (8.910) | -10.12 (6.555) | -8.38 (7.787) | -11.28 (8.998) | -12.04 (8.132) | -11.59 (10.112) | -12.18 (9.905) | -14.03 (9.425) | -12.54 (8.893) | -15.12 (8.437) | -13.87 (12.997) | -15.02 (9.197)

10. Secondary Outcome: Change From Baseline to Week 6 in Mean SBP and DBP Measured at Night by 24hr ABPM
Description: Mean changes from Baseline to Week 6 in DBP and SBP measured by 24hr ABPM at the end of up-titration recorded in the night. The night-time assessment period started at the time of the first reading at or after 6 pm and ended immediately before 6 am on the following day.
Time Frame: Night BP, Baseline, Week 6
Population: : ABPM Population with LOCF: This comprised all randomized subjects with efficacy (vital signs) data after a minimum of 2 weeks on treatment with valid Baseline and on-therapy ABPM measures. All efficacy data derived from ABPM assessments were summarized by this population
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lisinopril 10 | Lisinopril 20 | Lisinopril 40 | Carvedilol Controlled Release 20 | Carvedilol Controlled Release 40 | Carvedilol Controlled Release 80 | Carvedilol Controlled Release 20 Lisinopril 10 | Carvedilol Controlled Release 20 Lisinopril 20 | Carvedilol Controlled Release 20 Lisinopril 40 | Carvedilol Controlled Release 40 Lisinopril 10 | Carvedilol Controlled Release 40 Lisinopril 20 | Carvedilol Controlled Release 40 Lisinopril 40 | Carvedilol Controlled Release 80 Lisinopril 10 | Carvedilol Controlled Release 80 Lisinopril 20 | Carvedilol Controlled Release 80 Lisinopril 40
Number analyzed (Participants) | 29 | 30 | 38 | 27 | 34 | 33 | 35 | 37 | 34 | 32 | 35 | 34 | 28 | 33 | 34
mmHg
  Change in Night SBP from Baseline to Week 6 | -9.01 (10.635) | -11.58 (16.103) | -10.38 (8.600) | -4.28 (8.018) | -7.70 (10.178) | -7.71 (9.627) | -10.37 (11.517) | -9.94 (11.220) | -12.64 (11.301) | -10.02 (10.256) | -11.87 (12.031) | -11.25 (11.462) | -12.08 (9.486) | -14.12 (12.151) | -13.06 (10.651)
  Change in Night DBP from Baseline to Week 6 | -5.83 (6.602) | -6.78 (8.251) | -7.49 (6.085) | -3.20 (5.340) | -6.49 (5.723) | -5.34 (7.187) | -8.11 (7.260) | -7.03 (6.853) | -9.36 (7.068) | -8.23 (7.458) | -9.34 (8.960) | -9.09 (7.321) | -8.27 (6.002) | -9.88 (8.161) | -10.14 (7.468)

11. Secondary Outcome: Change From Baseline to Week 6 in Mean Trough Sitting SBP and Sitting DBP by Cuff Assessment
Description: Analysis of Change from Baseline to Week 6 in Mean sSBP and sDBP by Cuff Assessments at Drug Trough (20-24 hr) at End of Treatment Titration
Time Frame: Baseline, Week 6
Population: ITTE with LOCF. Intent to Treat Efficacy population is defined as all randomized subjects with efficacy (vital signs) data after a minimum of 2 weeks on treatment.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Lisinopril 10 | Lisinopril 20 | Lisinopril 40 | Carvedilol Controlled Release 20 | Carvedilol Controlled Release 40 | Carvedilol Controlled Release 80 | Carvedilol Controlled Release 20 Lisinopril 10 | Carvedilol Controlled Release 20 Lisinopril 20 | Carvedilol Controlled Release 20 Lisinopril 40 | Carvedilol Controlled Release 40 Lisinopril 10 | Carvedilol Controlled Release 40 Lisinopril 20 | Carvedilol Controlled Release 40 Lisinopril 40 | Carvedilol Controlled Release 80 Lisinopril 10 | Carvedilol Controlled Release 80 Lisinopril 20 | Carvedilol Controlled Release 80 Lisinopril 40
Number analyzed (Participants) | 42 | 41 | 42 | 40 | 40 | 40 | 41 | 42 | 43 | 42 | 43 | 40 | 39 | 43 | 41
mmHg
  Change in sSBP by Cuff from Baseline to Week 6 | -11.97 (13.671) | -10.85 (12.975) | -13.09 (10.200) | -5.68 (10.074) | -5.07 (15.610) | -8.88 (15.179) | -9.54 (14.373) | -11.84 (16.943) | -13.43 (15.279) | -9.79 (14.481) | -11.26 (15.056) | -13.49 (17.626) | -6.42 (16.409) | -9.00 (14.541) | -14.58 (16.176)
  Change in sDBP by Cuff from Baseline to Week 6 | -7.45 (13.671) | -5.32 (8.969) | -10.35 (7.627) | -6.87 (5.671) | -5.70 (9.760) | -7.54 (8.469) | -5.66 (8.949) | -10.02 (10.384) | -10.28 (8.543) | -8.73 (10.771) | -10.89 (10.757) | -9.63 (11.073) | -8.22 (9.203) | -9.45 (11.204) | -10.95 (8.624)

12. Secondary Outcome: Diastolic Responders, Defined as ≥ 10 mmHg Sitting (s)DBP Reduction From Baseline or a sDBP of <90 / 80 Millimeters (mm) of Mercury (Hg) for Non Diabetic / Diabetic Subjects Respectively (Based on Cuff Trough Measures)
Time Frame: Week 6
Population: as for outcome 11
Measure: Number; unit: participants
Arm/Group | Lisinopril 10 | Lisinopril 20 | Lisinopril 40 | Carvedilol Controlled Release 20 | Carvedilol Controlled Release 40 | Carvedilol Controlled Release 80 | Carvedilol Controlled Release 20 Lisinopril 10 | Carvedilol Controlled Release 20 Lisinopril 20 | Carvedilol Controlled Release 20 Lisinopril 40 | Carvedilol Controlled Release 40 Lisinopril 10 | Carvedilol Controlled Release 40 Lisinopril 20 | Carvedilol Controlled Release 40 Lisinopril 40 | Carvedilol Controlled Release 80 Lisinopril 10 | Carvedilol Controlled Release 80 Lisinopril 20 | Carvedilol Controlled Release 80 Lisinopril 40
Number analyzed (Participants) | 42 | 41 | 42 | 40 | 40 | 40 | 41 | 42 | 43 | 42 | 43 | 40 | 39 | 43 | 41
participants | 22 | 23 | 27 | 20 | 18 | 17 | 20 | 28 | 25 | 30 | 22 | 27 | 28 | 24 | 28

ADVERSE EVENTS:
Description: SAE/AE summary is based on the safety population, which comprised all randomized participants who received at least one dose of study medication; thus, the number of participants at risk differs by 1 for the Lis 20, Carv 40, Carv 40/Lis 40, and Carv 80/40 groups between the AE/SAE summary and the Participant Flow (all randomized participants).
Arm/Group | Lisinopril 10 | Lisinopril 20 | Lisinopril 40 | Carvedilol Controlled Release 20 | Carvedilol Controlled Release 40 | Carvedilol Controlled Release 80 | Carvedilol Controlled Release 20 Lisinopril 10 | Carvedilol Controlled Release 20 Lisinopril 20 | Carvedilol Controlled Release 20 Lisinopril 40 | Carvedilol Controlled Release 40 Lisinopril 10 | Carvedilol Controlled Release 40 Lisinopril 20 | Carvedilol Controlled Release 40 Lisinopril 40 | Carvedilol Controlled Release 80 Lisinopril 10 | Carvedilol Controlled Release 80 Lisinopril 20 | Carvedilol Controlled Release 80 Lisinopril 40
Serious Adverse Events (participants affected / at risk) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 1 | 3 | 0 | 1 | 1 | 1
Other Adverse Events (participants affected / at risk) | 22 | 15 | 21 | 20 | 17 | 13 | 19 | 20 | 30 | 21 | 33 | 19 | 13 | 38 | 15
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Lisinopril 10 | Lisinopril 20 | Lisinopril 40 | Carvedilol Controlled Release 20 | Carvedilol Controlled Release 40 | Carvedilol Controlled Release 80 | Carvedilol Controlled Release 20 Lisinopril 10 | Carvedilol Controlled Release 20 Lisinopril 20 | Carvedilol Controlled Release 20 Lisinopril 40 | Carvedilol Controlled Release 40 Lisinopril 10 | Carvedilol Controlled Release 40 Lisinopril 20 | Carvedilol Controlled Release 40 Lisinopril 40 | Carvedilol Controlled Release 80 Lisinopril 10 | Carvedilol Controlled Release 80 Lisinopril 20 | Carvedilol Controlled Release 80 Lisinopril 40
Abdominal pain (Gastrointestinal disorders) | 0/44 | 0/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 0/44 | 0/42 | 1/44 | 0/44 | 0/42
Alcoholism (Psychiatric disorders) | 0/44 | 0/42 | 0/43 | 1/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42
Anaemia (Blood and lymphatic system disorders) | 0/44 | 0/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 1/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42
Angioedema (Skin and subcutaneous tissue disorders) | 0/44 | 0/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 1/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42
Blood pressure increased (Investigations) | 0/44 | 0/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 0/44 | 0/42 | 1/44 | 0/44 | 0/42
Cardiac failure congestive (Cardiac disorders) | 0/44 | 0/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 1/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42
Cervical vertebral fracture (C2) (Injury, poisoning and procedural complications) | 0/44 | 0/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 0/44 | 0/42 | 0/44 | 1/44 | 0/42
Chest pain (General disorders) | 0/44 | 0/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 1/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42
Depression (Psychiatric disorders) | 0/44 | 0/42 | 0/43 | 1/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42
Drug abuse (Psychiatric disorders) | 0/44 | 0/42 | 0/43 | 1/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42
Gastritis (Gastrointestinal disorders) | 0/44 | 0/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 0/44 | 0/42 | 1/44 | 0/44 | 0/42
Headache (Nervous system disorders) | 0/44 | 0/42 | 0/43 | 1/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0/44 | 1/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42
Hypertension (worsening) (Vascular disorders) | 0/44 | 0/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 1/42
Ischaemic cerebral infarction (Nervous system disorders) | 0/44 | 0/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 1/43 | 0/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42
Left bundle branch block (Cardiac disorders) | 0/44 | 0/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 1/44 | 0/42 | 0/44 | 0/44 | 0/42
Lethargy (Nervous system disorders) | 0/44 | 1/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42
Listless (Psychiatric disorders) | 0/44 | 1/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42
Myocardial infarction (Cardiac disorders) | 0/44 | 0/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 1/44 | 0/42 | 0/44 | 0/44 | 0/42
Nausea (Gastrointestinal disorders) | 0/44 | 1/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42
Non-cardiac chest pain (General disorders) | 0/44 | 0/42 | 0/43 | 1/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42
Rib fracture (Injury, poisoning and procedural complications) | 0/44 | 0/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 1/44 | 0/42 | 0/44 | 0/44 | 0/42
Vaginal haemorrhage (Reproductive system and breast disorders) | 0/44 | 0/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 1/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Lisinopril 10 | Lisinopril 20 | Lisinopril 40 | Carvedilol Controlled Release 20 | Carvedilol Controlled Release 40 | Carvedilol Controlled Release 80 | Carvedilol Controlled Release 20 Lisinopril 10 | Carvedilol Controlled Release 20 Lisinopril 20 | Carvedilol Controlled Release 20 Lisinopril 40 | Carvedilol Controlled Release 40 Lisinopril 10 | Carvedilol Controlled Release 40 Lisinopril 20 | Carvedilol Controlled Release 40 Lisinopril 40 | Carvedilol Controlled Release 80 Lisinopril 10 | Carvedilol Controlled Release 80 Lisinopril 20 | Carvedilol Controlled Release 80 Lisinopril 40
Headache (Nervous system disorders) | 4/44 | 1/42 | 7/43 | 7/43 | 5/43 | 4/44 | 4/44 | 4/43 | 5/44 | 3/44 | 3/44 | 1/42 | 2/44 | 7/44 | 2/42
Dizziness (Nervous system disorders) | 3/44 | 3/42 | 3/43 | 3/43 | 4/43 | 3/44 | 1/44 | 3/43 | 6/44 | 3/44 | 5/44 | 3/42 | 2/44 | 4/44 | 0/42
Cough (Respiratory, thoracic and mediastinal disorders) | 6/44 | 3/42 | 1/43 | 1/43 | 0/43 | 0/44 | 2/44 | 2/43 | 4/44 | 2/44 | 7/44 | 5/42 | 1/44 | 2/44 | 2/42
Fatigue (General disorders) | 1/44 | 3/42 | 1/43 | 1/43 | 3/43 | 2/44 | 1/44 | 2/43 | 1/44 | 3/44 | 4/44 | 3/42 | 2/44 | 7/44 | 2/42
Nausea (Gastrointestinal disorders) | 3/44 | 1/42 | 1/43 | 3/43 | 2/43 | 0/44 | 2/44 | 3/43 | 1/44 | 1/44 | 2/44 | 0/42 | 1/44 | 3/44 | 0/42
Diarrhoea (Gastrointestinal disorders) | 1/44 | 2/42 | 0/43 | 1/43 | 0/43 | 0/44 | 1/44 | 1/43 | 2/44 | 3/44 | 2/44 | 2/42 | 1/44 | 4/44 | 1/42
Upper respiratory tract infection (Infections and infestations) | 3/44 | 0/42 | 2/43 | 0/43 | 0/43 | 0/44 | 3/44 | 1/43 | 5/44 | 1/44 | 1/44 | 1/42 | 1/44 | 0/44 | 1/42
Back Pain (Musculoskeletal and connective tissue disorders) | 0/44 | 1/42 | 0/43 | 2/43 | 1/43 | 1/44 | 0/44 | 1/43 | 1/44 | 2/44 | 3/44 | 0/42 | 2/44 | 2/44 | 0/42
Nasopharyngitis (Infections and infestations) | 0/44 | 1/42 | 1/43 | 1/43 | 0/43 | 1/44 | 1/44 | 0/43 | 1/44 | 1/44 | 3/44 | 1/42 | 0/44 | 1/44 | 3/42
Influenza (Infections and infestations) | 0/44 | 0/42 | 1/43 | 0/43 | 0/43 | 0/44 | 1/44 | 0/43 | 0/44 | 2/44 | 2/44 | 1/42 | 1/44 | 3/44 | 0/42
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0/44 | 0/42 | 1/43 | 0/43 | 1/43 | 1/44 | 0/44 | 0/43 | 0/44 | 0/44 | 1/44 | 1/42 | 0/44 | 0/44 | 3/42
Sinusitis (Infections and infestations) | 0/44 | 0/42 | 0/43 | 1/43 | 1/43 | 0/44 | 0/44 | 0/43 | 0/44 | 0/44 | 0/44 | 0/42 | 0/44 | 5/44 | 0/42
Myalgia (Musculoskeletal and connective tissue disorders) | 1/44 | 0/42 | 2/43 | 0/43 | 0/43 | 0/44 | 0/44 | 0/43 | 4/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0/44 | 0/42 | 1/43 | 0/43 | 0/43 | 1/44 | 3/44 | 0/43 | 0/44 | 0/44 | 0/44 | 1/42 | 0/44 | 0/44 | 1/42
Vertigo (Ear and labyrinth disorders) | 0/44 | 0/42 | 0/43 | 0/43 | 0/43 | 0/44 | 0/44 | 3/43 | 0/44 | 0/44 | 0/44 | 0/42 | 0/44 | 0/44 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the Publication of results from all centers of a multi-center trial but requests that reports based on Single-site data not precede the primary publication of the entire clinical trial.